CLINICAL TRIAL: NCT03019510
Title: Dawn Phenomena: Lowering Impaired Fasting Glucose Levels With Exercise (LIFE)
Brief Title: Lowering Impaired Fasting Glucose Levels With Exercise
Acronym: LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1202202 LIFE
Record Dates: First submitted 2016-12-19; First posted 2017-01-12 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- no exercise (Placebo Comparator): Subjects will be studied from 6 pm to 7 am following 48 hr of no exercise
  Interventions: Behavioral: No exercise; Behavioral: Morning exercise; Behavioral: Evening exercise
- morning exercise (Active Comparator): Subjects will be studied from 6 pm to 7 am. Subjects will have exercised at 7 am on that day.
  Interventions: Behavioral: No exercise; Behavioral: Morning exercise; Behavioral: Evening exercise
- evening exercise (Active Comparator): Subjects will be studied from 6 pm to 7 am. Subjects will exercise at 8 pm following dinner on the study day.
  Interventions: Behavioral: No exercise; Behavioral: Morning exercise; Behavioral: Evening exercise

INTERVENTIONS:
Behavioral: No exercise — No exercise will be done on the day of the study night to be tested
Behavioral: Morning exercise — Early morning exercise will be done on the day of the study night to be tested
Behavioral: Evening exercise — Evening exercise will be done on the day of the study night to be tested

SUMMARY:
Morning hyperglycemia plays a role in the future development of insulin resistance and type 2 diabetes (T2D) (8) and is associated with numerous microvascular and cardiovascular complications and renal disease. These augmented morning glucose levels are due to an elevated endogenous glucose production (EGP), as a result of a loss of coordination between glucose levels and insulin secretion, and possibly hyperglucagonemia during the overnight period. Exercise stimulates glucose uptake and increases insulin sensitivity acutely, and may be the best lifestyle intervention to minimize the nocturnal rise in glucose levels. Prescription of the timing of exercise relative to a meal and/or to the overnight period may be particularly critical for individuals that have impaired fasting glucose (IFG) levels. Surprisingly little is known about the overnight period when elevated EGP and the synchrony between glucose and c-peptide/glucagon levels becomes disturbed. This novel study will provide insight into the hormonal/metabolic milieu of a dinner meal, the evening and overnight period that occurs in non-obese, OB and OB+IFG individuals; it will also establish if the timing of exercise can attenuate nocturnal glucose elevations, and if this is associated with improved hormonal synchrony. This project will compare EGP, β-cell function and hormonal responses between morning and evening exercise on the postprandial and overnight period in obese individuals with/without IFG levels. Fifty-four subjects will be studied during the evening meal (EGP and β-cell function), postprandially and through the overnight period (1600-0700 h), allowing us to examine some of the potential mechanisms for the elevation in overnight glucose levels. This is the first study that will examine this issue from pre-dinner through the night while previous studies have only examined chronically fasted individuals and this study will lay the groundwork for understanding the pathology of the predawn phenomena in OB+IFG individuals. These potentially translational findings may impact the efficiency of physician communication to patients concerning exercise. These investigators are one of the few groups that study subjects through the overnight period and have the facilities and capability to do this research.

DETAILED DESCRIPTION:
In individuals with type 2 diabetes (T2D), chronically elevated glucose and insulin levels result in numerous health complications. Maintaining tight glucose control is difficult for individuals with T2D, particularly in the postprandial period and in the morning period just prior to waking. In the postprandial period, the combined effect of insulin resistance and beta cell dysfunction results in a prolonged elevation in glucose levels, and augmented insulin levels in an attempt to reduce the circulating glucose levels. In the overnight period, there is evidence of enhanced endogenous glucose production and of a disruption of the interaction between glucose levels and insulin secretion. Early work in individuals with T2D demonstrated that with continued fasting, glucose levels stopped declining in the evening and subsequently rose throughout the night to reach a morning maximum, and this elevation persisted till noon. Additionally these authors demonstrated that insulin levels and insulin secretion rates did not parallel the nocturnal glucose changes in individuals with T2D, while in the controls the nocturnal glucose and insulin secretion rates coincided. Evidence is also emerging that hyperglucagonemia may be occurring in the setting of deficient insulin secretion, and may be playing a role in the elevated postprandial glucose levels and in the overnight period. These studies provide preliminary evidence that there is disruption in the fine coordination between glucose levels and glucagon and insulin secretion, and that this is exacerbated more in the overnight period than during the waking hours. Previous studies examining the overnight period have been conducted following prolonged fasting (~24-34 h), however, most people do not fast for extended periods of time prior to going to bed. Additionally, individuals with T2D often know that meal composition the evening prior can exacerbate the elevated fasting glucose levels the following morning, thus highlighting the need to examine the effect of meal composition on overnight glucose control. To date, very little is known about the pathology of why fasting glucose levels are elevated in many obese individuals. There appears to be asynchrony between glucose and insulin levels in the overnight period but very little research has focused on this phenomenon or how meal composition affects overnight glucose levels. This study will provide evidence of potential mechanisms for the elevation in overnight glucose levels and the findings will be translatable for individuals with impaired fasting glucose (IFG) levels to understand the importance of meal composition in the evening period.

The specific aims of this project are:

1. To examine the hormonal responses (glucagon, c-peptide, insulin, incretins) in response to a meal in the postprandial period and the synchronization between glucose and insulin/glucagon during the overnight period in non-obese individuals and obese individuals with impaired fasting glucose levels (IFG).
2. To determine if the meal composition (standard meal: 55% carbohydrate, 20% protein, 25% fat vs. high fat/fructose: 40% carbohydrate- 25% fructose, 40% fat, 20% protein) will alter the hormonal responses (glucagon, insulin, incretin) in the postprandial period, and if this change in meal composition will impact glucagon levels and glucose/c-peptide synchrony in the overnight period.

Experimental design: Subjects will participate three times; 1) no exercise, 2) 2 hr post dinner exercise, and 3) morning exercise (~7am). The order in which subjects undergo each treatment will be randomized prior to study enrollment. Eligible subjects will initially undergo baseline testing for assessment of body composition, exercise stress test and blood screening. All subjects will have impaired fasting glucose levels. All subjects will undergo 3 study days that will start at ~1600 h and continue until 0700 h the following morning. They will receive a standard meal (55% carbohydrate, 20% protein, 25% fat) at 1800 h and blood samples will be taken from ~4:30 pm until 7 am.

ELIGIBILITY:
Inclusion Criteria:

25-65 yrs of age body mass index (BMI): 30-45 kg/m2 for the obese subjects <24.5 kg/m2 for the non-obese subjects weight stable during prior 6 months non-smokers OB with impaired fasting glucose: elevated elevated morning fasting glucose levels >110 mg/dL for 5 of 7 days non-obese and OB subjects: fasting glucose levels < 100 mg/dL - 2hr OGTT glucose value <140 mg/dL

Exclusion criteria overt cardiovascular disease sleep apnea surgical history for weight loss use of weight-loss medications or active dieting participate in exercise > 3 days/wk per week at a moderate or vigorous intensity pregnant or lactating women. Medications for glycemic control (including insulin), β-blockers, glucocorticoids, testosterone, or other medications for chronic pulmonary, cardiac or other systemic diseases.

Significant hypertension BP > 180 systolic or > 100 diastolic, at rest. Untreated hypothyroidism or hyperthyroidism (will be included if treated and euthyroid) Active users of tobacco and chronic alcohol abuse. Renal, hepatic, pulmonary, adrenal, or pituitary disease. Liver function tests with > 2xULN.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-10; Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
fasting glucose level | avg of every 15 min for 1 hr will be compared between interventions
  the hour prior to study completion will be used for this measurement

SECONDARY OUTCOMES:
endogenous glucose production | the endogenous glucose production for 4 hr will be compared between intervention
insulin concentrations | the insulin concentrations 13 hr will be compared between interventions
glucagon concentrations | the glucagon concentrations for 13 hr will be compared between interventions
beta cell function | beta cell function determined for 4 hr postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No